CLINICAL TRIAL: NCT00957645
Title: Central Post-Stroke Pain - a Prospective Study of Consecutively Admitted Patients With Recent Stroke
Brief Title: Central Post-Stroke Pain - a Prospective Study
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20060116
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pain
Keywords: Central post-stroke pain; post-stroke pain; shoulder pain
MeSH Terms: conditions — Pain; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Part 1: The purpose of the first part of the study is to investigate the prevalence of pain at stroke onset and 3 and 6 months after stroke in a consecutive cohort of stroke patients admitted to a stroke unit.

Part 2: The purpose of the second part of the study is to identify patients who develop central post-stroke pain within the first 6 months following stroke and to try to identify early prognostic factors for the development of pain.

DETAILED DESCRIPTION:
Part 1:

* Within 3 days of admission: medical history, pain history, sensory examination
* Telephone follow-up at 3 and 6 months post-stroke: pain history

Part 2:

* Medical history, Pain history, Sensory examination

ELIGIBILITY:
Inclusion Criteria:

* Recent cerebrovascular stroke

Exclusion Criteria:

* Severe dementia, aphasia or psychosis
* Patients who cannot cooperate at time of inclusion
* Patients who do not understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive stroke patients admitted to the Stroke Unit of the Department of Neurology at Aarhus University Hospital between February 2008 to October 2009
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Klit, MD, Principal Investigator — Danish Pain Research Center